CLINICAL TRIAL: NCT03247166
Title: A Study to Evaluate the Safety and Effectiveness of the TOPS™ SP System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-36-17
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower Back and Leg Pain Patients (Experimental): Patients suffering from lower back and leg pain resulting in degenerative spondylolisthesis and/or spinal stenosis will undergo treatment using the TOPS™ System
  Interventions: Device: TOPS™ System

INTERVENTIONS:
Device: TOPS™ System — The TOPS™ System is an alternative to spinal fusion that is designed to stabilize but not fuse the effected vertebrai level to alleviate pain stemming from degenerative joints

SUMMARY:
The TOPS™ SP System is intended to provide stabilization in skeletally mature patients. The system is designed to afford motion of the spine segment without fusion. The pur0pose of this prospective clinical study is to establish the safety and effectiveness of the TOPS™ System, when used following decompression, in the treatment of lower back and sciatic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic monosegmental lumbar spinal stenosis or facet arthrosis
* Patients with degenerative spondylolisthesis
* Patients with at least 3 months failed conservative treatment
* Narrowing of the lumbar spinal canal
* Patients with lower back pain or sciatica

Exclusion Criteria:

* Discogenic back pain at TOPS System level
* Back or non-radicular leg pain of unknown etiology at TOPS System level
* Lytic spondylolisthesis at TOPS System level
* More than one motion segment involved in degenerative pathology to the extent that justifies its inclusion in the surgical procedure
* Known allergy to titanium and/or polyurethane

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pain Improvement | 24 months
  Subjects having a 15% reduction in the Oswestry Low Back Pain Disability Questionnaire score as compared to their preoperative Oswestry score
Function Improvement | 24 months
  Subjects having a 15% reduction in the Oswestry Low Back Pain Disability Questionnaire score as compared to their preoperative Oswestry score
Fusion Prevention | 24 months
  The subjects will be considered a failure if fusion occurs as defined in the radiographic protocol

OTHER OUTCOMES:
Safety | 24 months
  Subjects with no serious device complications as defined in the radiological protocol

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Behrbalk, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No